CLINICAL TRIAL: NCT06817798
Title: Effects of Specific Foot Mobility Techniques on Biomechanical and Functional Parameters in Young Adults: A Randomized Controlled Trial
Brief Title: Impact of Foot Mobility Techniques on Balance and Pressure in Young Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cooperativa de Ensino Superior, Politécnico e Universitário (Other)
Responsible Party: Principal Investigator, Maria Paço, Principal investigator, Cooperativa de Ensino Superior, Politécnico e Universitário
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Foot mobility_2025
Record Dates: First submitted 2025-01-22; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Foot Mobility; physiotherapy; biomechanics; balance; plantar pressure; baropodometry; manual therapy; lower limb function; rehabilitation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specific foot mobility (Experimental): Specific mobility of the foot, performed bilaterally.
  Interventions: Other: Specific foot mobility
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Specific foot mobility — Specific mobility of the foot, performed bilaterally.
  Arms: Specific foot mobility

SUMMARY:
This study aims to evaluate the effectiveness of specific foot mobility techniques on functional and biomechanical parameters of the foot in young adults aged 18 to 24 years. The study employs a randomized controlled trial design with the following key components:

Key outcomes include:

Baropodometric pressures (measured using a baropodometric platform). Balance (evaluated through the Y-Balance Test). Navicular height (assessed using the Navicular Drop Test) Anterior functional reach (measured through functional reach test)

DETAILED DESCRIPTION:
This study explores the immediate and short-term effects of specific foot mobility techniques on functional and biomechanical outcomes in healthy young adults. The research is grounded in the growing recognition of the foot's critical role in postural control, balance, and lower-limb biomechanics.

The intervention consists of foot mobility techniques designed to improve joint mobility and overall foot function. These techniques will be applied bilaterally. The study employs a randomized controlled trial design, with participants randomly allocated to either the experimental group (receiving the intervention) or the control group (receiving no treatment during the intervention period).

Participants are assessed at three time points:

Baseline (M0): Before the intervention. Immediately Post-Intervention (M1). Follow-Up (M2): 24 hours after the intervention.

The primary outcomes include:

Changes in plantar pressure distribution and postural control as measured by a baropodometric platform.

Balance performance assessed through the Y-Balance Test. Navicular height variation evaluated using the Navicular Drop Test. Anterior functional reach, measured by Functional Reach Test. The study focuses on identifying measurable improvements in functional and biomechanical parameters that may enhance clinical approaches to foot health and rehabilitation. By targeting a young and healthy population, the research aims to establish a foundation for further studies in other age groups and clinical conditions. This work aims to contribute to evidence-based practices in manual therapy and foot biomechanics.

ELIGIBILITY:
Inclusion Criteria:

* minimum age of 18 years.

Exclusion Criteria:

* pregnant women,
* individuals with lesions in the lower limbs in the last 12 months,
* history of congenital deformity in the lower limb
* presence of vestibular or balance disorders
* users of corrective insoles or orthoses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Balance - Y balance test | M0: Before intervention; M1: Immediately after intervention; M2: 24h after intervention.
  Assesses dynamic balance by having participants reach as far as possible in multiple directions with one foot while maintaining balance on the other, providing insight into lower limb stability and control.
Baropodometric pressure | M0: Before intervention; M1: Immediately after intervention; M2: 24h after intervention.
  To assess load distribution, participants will be instructed to stand on the force platform in an orthostatic position for 30 seconds.
Navicular height - Navicular drop test | M0: Before intervention; M1: Immediately after intervention; M2: 24h after intervention.
  The navicular drop test will be performed. In this test, the height of the navicular bone is measured with a caliper (in millimetres) from the ground to the most distal point of this bone.
Anterior functional reach - functional reach test | M0: Before intervention; M1: Immediately after intervention; M2: 24h after intervention.
  The participant is instructed to stand close to, but not touching, a wall and position the arm that is closer to the wall at 90 degrees of shoulder flexion with a closed fist. The assessor records the starting position at the 3rd metacarpal head on the yardstick. Then, the participant is instructed to "Reach as far as you can forward without taking a step." The location of the 3rd metacarpal is then recorded in this position. The difference between the start and end position is the reach distance.

CONTACTS AND LOCATIONS:
Locations (1):
- Escola Superior de Saúde do Vale do Ave, Vila Nova de Famalicão, Braga District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
eciding whether to share Individual Participant Data (IPD) involves weighing several considerations... we have to further reflect to make an informed decision about sharing IPD, balancing the potential benefits to the scientific community with the responsibility to protect participant rights and data integrity.